CLINICAL TRIAL: NCT01017198
Title: An Assessment of the Effect of Food and Antacid on BIIB021 Pharmacokinetics in Subjects With Advanced Solid Tumors.
Brief Title: Effect of Food and Antacid on BIIB021 With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 120ST104
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2011-01

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — 6-chloro-9-(4-methoxy-3,5-dimethylpyridin-2-ylmethyl)-9H-purin-2-ylamine; Food; Antacids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BIIB021 and Food (Experimental): The food phase will assess the effect of a high fat meal on the pharmacokinetics of BIIB021.
  Interventions: Drug: BIIB021 and Food
- BIIB021 and Antacid (Experimental): Antacid phase will assess the effect of an antacid on the pharmacokinetics of BIIB021.
  Interventions: Drug: BIIB0121 and Antacid

INTERVENTIONS:
Drug: BIIB021 and Food — Assessing the effect of food use on BIIB021
  Arms: BIIB021 and Food
Drug: BIIB0121 and Antacid — Assessing the effect of antacid use on BIIB021
  Arms: BIIB021 and Antacid

SUMMARY:
This study is designed to assess the effect of food and antacid use on the pharmacokinetic properties of BIIB021.

DETAILED DESCRIPTION:
This study has 2 phases (the Food Phase and the Antacid Phase), each consisting of a 2-period, 2-sequence, 2-treatment crossover design. The Food Phase will assess the effect of a high fat meal on the pharmacokinetics of 100 mg BIIB021, and the Antacid Phase will assess the effect of an antacid (ranitidine) on the pharmacokinetics of 450 mg BIIB021 in the same subjects. Ranitidine 150 mg will be taken the evening before and the morning of the antacid dosing day.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically confirmed solid tumors who have failed or are not candidates for standard therapies or for whom no approved therapy is available.
* Eastern Cooperative Oncology Group (ECOG) performance status of greater or equal to 2.
* Medically able to tolerate a high fat meal and to fast as per protocol.
* Expected survival time of at least 3 months in the opinion of the Investigator.
* Ability to take ranitidine as per protocol.
* Must be able to swallow and retain oral medication.
* Lab values consistent with adequate renal, hepatic, and bone marrow functions.
* Electrocardiogram (ECG) with QTc of ≤450 msec for men or ≤470 msec for women and no clinically significant findings.

Exclusion Criteria:

* Pregnant (positive pregnancy test) or nursing women.
* Previous treatment with an Hsp90 inhibitor.
* Use of antacids within 7 days of Study Day 1.
* Prior antitumor therapies, including prior experimental agents or approved antitumor therapies within 28 days of the first dose of BIIB021.
* Major surgery or radiation within 28 days of the first dose of BIIB021.
* Uncontrolled, severe medical illness, which in the opinion of the Investigator and/or Sponsor could compromise protocol objectives.
* History of gastrectomy or major surgery to small intestine.
* History of exocrine pancreatic insufficiency.
* Chronic diarrhea (excess of 2 to 3 stools/day above normal frequency).
* Active bacterial or viral infection requiring concurrent treatment.
* History of hepatitis B or C or human immunodeficiency virus.
* History of central nervous system metastasis.
* Any thrombotic event occurred <3 months prior to Day 1.
* Conditions that may predispose subjects to seizures: History of seizure, previous significant head trauma
* Drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to assess the pharmacokinetics of BIIB021 taken under fed conditions compared to BIIB021 taken under fasting conditions in subjects with advanced solid tumors. | Cycle 1, Day 3

SECONDARY OUTCOMES:
To assess the pharmacokinetics of BIIB021 taken with an antacid (ranitidine) compared to BIIB021 taken with no antacid, both under fasting conditions | Cycle 1, Day 8 and Day 10
To evaluate the safety and tolerability of BIIB021 | 6 months
To evaluate the antitumor activity of BIIB021 | 6 months
To evaluate the effect of BIIB021 on pharmacodynamic biomarkers. | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Reseach Facility, Scottsdale, Arizona
  - Reseach Facility, Encinitas, California
  - Reseach Facility, San Antonio, Texas